CLINICAL TRIAL: NCT05699603
Title: Phase IIA, Single-Arm, Open- Label, Clinical Trial of Calcipotriene Plus 5-fluorouracil Immunotherapy for Skin Cancer Prevention in Organ Transplant Recipients
Brief Title: Testing the Efficacy of Topical Calcipotriene Plus 5-Fluorouracil Combination to Activate the Immune System Against Precancerous Skin Lesions in Organ Transplant Recipients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2023-00310; P30CA023074 (NIH); UG1CA242596 (NIH); NCI-2023-00310 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002897 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ22-10-01 (Other: DCP)
Record Dates: First submitted 2023-01-25; First posted 2023-01-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Biopsy; calcipotriene; Fluorouracil; dehydroftorafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (calcipotriene, fluorouracil) (Experimental): Participants receive calcipotriene plus fluorouracil cream topically BID for 6 consecutive days on study. Participants also undergo skin biopsies throughout the study. Patients who continue to experience AKs at week 8 may receive a second course of calcipotriene plus fluorouracil cream topically BID for 6 consecutive days on study.
  Interventions: Procedure: Biopsy; Drug: Calcipotriene; Drug: Fluorouracil

INTERVENTIONS:
Procedure: Biopsy — Undergo skin biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Calcipotriene — Applied topically
  Other Names: Calcipotriol; Dovonex
Drug: Fluorouracil — Applied topically
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757

SUMMARY:
This phase IIA study evaluates the effects of calcipotriene plus 5- fluorouracil immunotherapy for skin cancer prevention in organ transplant recipients. Solid organ transplant recipients are at high risk of developing skin cancer. Actinic keratosis (AK), is a premalignant skin lesion that can progress to squamous cell skin cancer. In this study, solid organ transplant recipients with multiple AKs are treated with topical calcipotriene and 5-FU to evaluate how effective this therapy is against AKs and if this could lower their risk of skin cancer. Topical calcipotriene is a form of vitamin D and is used to treat psoriasis. Prior research reported immunomodulatory effects in the skin induced by topical calcipotriene. Topical 5- fluorouracil is a chemotherapy agent and is one of the therapy options for multiple AKs in specific clinical scenarios. Prior research indicates that topical calcipotriene used together with topical 5-FU was more effective in treating multiple AKs than 5-FU alone in individuals with healthy immune system. This study is investigating now if similar beneficial effects can be seen in immunosuppressed individuals who are solid organ transplant recipients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the induction of CD4+ TRM cells (CD3+CD4+CD103+) in the actinic keratosis at one day after completing one and two courses of calcipotriene plus 5-fluorouracil (5-FU) immunotherapy compared with before treatment.

SECONDARY OBJECTIVES:

I. To evaluate the persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK at 6 months after initiation of treatment compared with before treatment.

II. To evaluate the persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK at 6 months after initiation of treatment compared with after completing one and two courses of treatment.

III. To determine the percent reduction in the number of AKs on the treated areas at 8 weeks after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment.

IV. To determine the erythema extent and intensity scores of the treated anatomical sites at one day after the completion of one and two courses of calcipotriene plus 5-FU immunotherapy.

V. To determine differences in AK clearance between the treated anatomical sites (upper extremities versus [vs.] face vs. scalp).

VI. To assess the safety and tolerability of one and two courses of calcipotriene plus 5-FU treatment.

VII. To assess any incidence of biopsy-proven acute organ rejection of the graft.

EXPLORATORY OBJECTIVES:

I. To determine the percentage of participants with a new diagnosis of squamous cell carcinoma (SCC) on the treated anatomical sites at 6 months after the initiation of treatment compared with the identical duration prior to therapy.

II. To evaluate the persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK at 8 weeks after treatment with one and two courses of calcipotriene plus 5-FU compared with before treatment.

III. To evaluate the induction of TSLP, CD8+ TRM and natural killer (NK) cell infiltrates in the AK at one day after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment.

IV. To evaluate the induction of other immune cells/factors in the AK at one day after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment.

V. To determine the induction of TSLP, CD3+ T, CD4+ T, CD8+ TRM, NK cell and other immune cells/factors in the AK at one day after two courses compared with one day after one course of calcipotriene plus 5-FU immunotherapy.

VI. To evaluate the persistence of CD8+ TRM, NK cells in the AK at 8 weeks after treatment with one and two courses of calcipotriene plus 5-FU compared with before treatment.

VII. To evaluate the persistence of CD8+ TRM, NK cells in the AK at 6 months after initiation of treatment compared with before treatment. VIII. To compare the immune infiltrate in any SCC that develops over 6 months after one and two courses calcipotriene plus 5-FU immunotherapy with SCCs that developed before treatment using archived tumor samples.

IX. To evaluate the effect of number and type of field therapy and the number of cryotherapies after the trial, age, gender, history of immunosuppressive therapy, exposure to ionizing radiation or chemical carcinogens before and after transplantation, genetic factors (Fitzpatrick skin type I, II and III), pre-transplantation end-organ disease on SCC outcomes in OTRs.

X. To compare the immune induction outcomes in AKs versus the normal skin samples.

OUTLINE:

Participants receive calcipotriene plus 5-fluorouracil cream topically twice a day (BID) for 6 consecutive days on study. Participants also undergo skin biopsies throughout the study. Patients who continue to experience AKs at week 8 may receive a second course of calcipotriene plus 5-fluorouracil cream topically BID for 6 consecutive days on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had received a kidney or lung transplant >= 2 years before enrollment in the study with a stable status of transplanted graft (participants must have visited their transplant specialist within 6 months before enrolling to the study, documenting stable graft safety). The target population includes patients who are on tacrolimus and/or MMF without voriconazole as their immunosuppressive regimen.
* Presence of four to fifteen clinically typical, visible, and discrete AKs in 25 cm^2 on any of the following anatomical sites: upper extremities, face, and/or scalp.
* Age of at least 18 years. Because no dosing or adverse event (AE) data are currently available on the use of calcipotriene plus 5-FU in participants <18 years of age, children and adolescents are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Karnofsky performance status >= 60%.
* Leukocytes >= 3,000/microliter and < 12000/ microliter.
* Absolute neutrophil count >= 1,000/microliter.
* Platelets >= 100,000/microliter.
* Creatinine =< 1.5 × institutional upper limit of normal.
* Baseline respiratory requirement for lung transplant recipients:

  * Respiratory rate within 12-18/min
  * PO2 saturation within 90-100mmHg
* Female participants must be non-reproductive potential (i.e., post-menopausal by a history of age > 50 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, history of bilateral tubal ligation, or history of bilateral oophorectomy) OR must have a negative urine pregnancy test. The effects of calcipotriene plus 5-FU on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because of unknown teratogenic effect, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Ability and willingness to participate in the study.

Exclusion Criteria:

* OTRs with any sign of organ rejection are not eligible.
* Patients who received any systemic cancer therapy or radiation within =< 1 year (y) of study enrollment, or have a diagnosis requiring them to receive such treatment(s) are excluded.
* Patients with known dihydropyrimidine dehydrogenase deficiency (due to the higher risk of 5-FU toxicity).
* Patients with known history of hypercalcemia or vitamin D toxicity.
* History of treatment with calcipotriene plus 5-FU within one year before enrollment in the study.
* The treatment area is within 5 cm of an incompletely healed wound or a suspected basal cell or squamous cell carcinoma.
* The treatment area contained hypertrophic and hyperkeratotic lesions, cutaneous horns, or lesions that had not responded to repeated cryotherapy.
* Participants may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to calcipotriene and or 5-FU
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because there is an unknown but potential risk for teratogenic or abortifacient effects. Also, there is unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with calcipotriene plus 5-FU, breastfeeding should be discontinued if the mother is treated.
* Participants who are HIV-positive will be excluded from the study. There is a higher risk of organ rejection in HIV-positive patients, and also a higher risk of developing skin cancer, related to their infection-associated immunosuppressed state and drug-induced immunosuppression for preventing organ rejection. In addition, considering HIV's adverse effects on CD4+ T cell function and the fact that the topical medication in this study is specifically designed to target CD4+ T cells, we plan to exclude HIV positive patients in order to avoid this confounding factor on the primary endpoint of the study.
* Participants with known history of chronic hepatitis B, or hepatitis C will be excluded from the study in order to avoid confounding an existing condition with an immune response to the study agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Induction of CD4+ TRM cells (CD3+CD4+CD103+) in the actinic keratosis | At one day after completing one and two courses of calcipotriene plus 5-FU immunotherapy
  Will be assessed at one day after completing one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment. Paired t test will be performed to evaluate whether the changes from baseline are significantly different from 0.

SECONDARY OUTCOMES:
Persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK | At 6 months
  Will be assessed after initiation of treatment compared with after initiation of treatment compared with before treatment. The mean change from baseline at 8 weeks and 6 months, respectively, after one and two courses and the associated 95% CI will be reported for both AK and normal skin.
Persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK | At 6 months
  Will be assessed after initiation of treatment compared with after completing one and two courses of treatment. The mean change from baseline at 8 weeks and 6 months, respectively, after one and two courses and the associated 95% CI will be reported for both AK and normal skin.
Percent reduction in the number of AKs | At 8 weeks
  Will be assessed on the treated areas at 8 weeks after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment.
Erythema extent and intensity scores of the treated anatomical sites | At one day after the completion of one and two courses
  Will be assessed at one day after the completion of one and two courses of calcipotriene plus 5-FU immunotherapy using the mean changes and the associated 95% CIs. The percentage of the participants with AK clearance (i.e., response to the treatment) and the exact (Clopper-Pearson) 95% CI will be reported by the treated anatomical sites.
Differences in AK clearance | At week 24
  Will be assessed between the treated anatomical sites (upper extremities vs. face vs. scalp).
Incidence of adverse events | After of one and two courses of calcipotriene plus 5-FU treatment
  Will be assessed after of one and two courses of calcipotriene plus 5-FU treatment.
Incidence of biopsy-proven acute organ rejection of the graft | At week 24
  The exact (Clopper-Pearson) 95% CI will be reported.

OTHER OUTCOMES:
Percentage of participants with new diagnosis of SCC on the treated anatomical sites | At 6 months
  Will be assessed after the initiation of treatment compared with the identical duration prior to therapy.
Persistence of CD4+ TRM (CD3+CD4+CD103+) in the AK | At 8 weeks
  Will be assessed after treatment with one and two courses of calcipotriene plus 5-FU compared with before treatment.
Induction of TSLP, CD8+ TRM and natural killer (NK) cell infiltrates in the AK | At one day after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment
Induction of other immune cells/factors in the AK | At one day after one and two courses of calcipotriene plus 5-FU immunotherapy compared with before treatment
Induction of TSLP, CD3+ T, CD4+ T, CD8+ TRM, NK cell and other immune cells/factors in the AK | At one day after one and two courses of calcipotriene plus 5-FU immunotherapy
Persistence of CD8+ TRM, NK cells in the AK | At 8 weeks
  Will be assessed after treatment with one and two courses of calcipotriene plus 5-FU compared with before treatment.
Persistence of CD8+ TRM, NK cells in the AK | At 6 months
  Will be assessed after initiation of treatment compared with before treatment.
Compare the immune infiltrate in any SCC | At 6 months
  Will be assessed after one and two courses calcipotriene plus 5-FU immunotherapy with SCCs that developed before treatment using archived tumor samples.
Effect of number and type of field therapy and the number of cryotherapies | Up to 2 years
  Will be assessed after the trial, age, gender, history of immunosuppressive therapy, exposure to ionizing radiation or chemical carcinogens before and after transplantation, genetic factors (Fitzpatrick skin type I, II and III), pre-transplantation end-organ disease on SCC outcomes in organ transplant recipients (OTRs).
Comparison of the immune induction outcomes in AKs versus the normal skin samples | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shadmehr Demehri, Principal Investigator — University of Arizona Cancer Center - Prevention Research Clinic
Locations (4):
- United States (4):
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm